CLINICAL TRIAL: NCT06876129
Title: Pharmacologic Augmentation of TMS for Depression With D-serine
Acronym: PAT-DS
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Joshua C. Brown, MD, PhD, Assistant Professor, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024P001927
Record Dates: First submitted 2024-08-12; First posted 2025-03-14 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: The proposed study is a randomized controlled trial with two groups: 1) placebo + TMS and 2) DS + TMS.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Subjects will be randomized into the placebo (n = 30) or D-serine group (n = 30) via a randomization list generated by the McLean Pharmacy to produce equal groups. The research pharmacist is the only one unblinded and will create the randomization table for the placebo and D-serine assignments. The study staff will then pick up the medications in a blinded state (e.g., bottles labeled "A" or "B"). Only at the end of the study will the pharmacy then reveal the drugs corresponding to the label. The placebo is sourced from the same pharmacy as D-serine and have been requested to be in identical capsules.
  Subjects will not be randomized into their TMS group and will either receive iTBS using our Magventure TMS device or 18-Hz H1 TMS using our dTMS Brainsway device. Subjects will have their TMS protocol/treatment determined at the time of consultation according to clinical appropriateness as is the standard of care at the TMS clinic at McLean Hospital.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo + TMS
  Interventions: Device: TMS
- D-serine (Active Comparator): D-serine + TMS
  Interventions: Combination Product: D-serine + TMS

INTERVENTIONS:
Device: TMS — Subjects will either receive iTBS using a Magventure TMS device or 18-Hz H1 TMS using a dTMS Brainsway device plus placebo.
  Arms: Placebo
Combination Product: D-serine + TMS — D-serine, 80 mg/kg, oral administration, will be advised to be taken 1-hour prior rTMS treatment day (Mon-Fri) for 6 weeks. Dosing is based on maximal plasticity at 80 mg/kg, and clinical dose-finding studies demonstrating that doses between 60 - 120 mg/kg were superior in clinical effectiveness to 30 mg/kg and were safe.
  Subjects will not be randomized into their TMS group and will either receive iTBS using a Magventure TMS device or 18-Hz H1 TMS using a dTMS Brainsway device. Subjects will have their TMS protocol/treatment determined at the time of consultation according to clinical appropriateness as is the standard of care at the TMS clinic at McLean Hospital.
  Arms: D-serine

SUMMARY:
The goal of this study is to test whether combining D-serine with 30 treatments of a) iTBS and b) 18-Hz protocols will enhance clinical outcomes compared to rTMS with placebo (i.e., sugar pill). The investigators hypothesize that NMDA receptor activation via D-serine combined with repeated sessions of rTMS will produce greater clinical outcomes than iTBS with placebo and 18-Hz with placebo.

DETAILED DESCRIPTION:
Consent Process:

After referral from the clinician, subjects will be contacted either by phone, by email, or in person, advised of the opportunity to participate in this study, and informed about what the study will entail. Subjects will give their own consent and will be over the age of 18.

Study Procedures:

All procedures may be available to all participants. If the participant agrees to take part in this study, the participant will be asked to undergo the following procedures during the experimental visit.

Clinical Measurement Initiative (CMI) Data: As part of routine clinical care, patients receiving TMS at McLean Hospital complete computerized clinician administered and patient self-reported assessments of clinical symptoms on admission and at interim and discharge points in their care. The computerized assessments are part of McLean Hospitals Clinical Measurement Initiative (CMI), which uses Research Electronic Data Capture (REDCap) software and a McLean-developed reporting module to generate individual patient reports used in ongoing clinical care and patient outcomes monitoring. The CMI was implemented in the McLean TMS program in May 2010. The investigators plan to conduct data analyses examining changes in TMS patient self-report of symptoms on the following standardized, validated surveys: Quick Inventory of Depressive Symptomatology Self Report (QIDS-SR) and Patient Health Questionnaire-9 (PHQ-9), Generalized Anxiety Disorder-7 which will be self-administered at treatment #1, #9, #14, #19, #24, #29, and #34, as well as clinician-administered Clinical Global Impression-Severity (CGI-S) at the point of consultation.

Transcranial Magnetic Stimulation (TMS): TMS involves a procedure where parts of the participant's brain will be non-invasively (i.e. indirectly) stimulated by magnetic pulses. Repetitive TMS (rTMS) administered in the study does not differ from standard of care as practiced in the McLean Clinic. Therefore, all patients will receive standard of care treatment combined along with either placebo or d-serine, designed to enhance clinical benefits.

Visits:

All visits follow our normal clinical schedule:

Visit 1: Participants will first undergo a TMS consultation to determine eligibility to safely receive TMS and assess clinical appropriateness for TMS.

Visit 2-37: 30 sessions of rTMS sessions (10-20 minutes long) daily, Mondays through Fridays, excluding weekends and holidays.

Drugs to be used (dose, method, schedule of administration, dose modifications, toxicities), include:

D-serine, 80 mg/kg (max 7g), oral administration, will be advised to be taken 1-hour prior rTMS treatment day (Mon-Fri) for 6 weeks. Dosing is based on maximal plasticity at 80 mg/kg, and clinical dose-finding studies demonstrating that doses between 60 - 120 mg/kg were superior in clinical effectiveness to 30 mg/kg and were safe. The drug will stopped at the discretion of the study clinicians after evaluation and assessment of any signs of adverse effects or signs of clinical worsening.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of MDD
* English-speaking
* Adults aged 18-80
* Must be able to swallow capsules

Relative contraindications/possible exclusion criteria:

* Containing any implanted metal or devices
* Current or previous seizure history
* Active substance use that may significantly alter the seizure threshold

Any further safety clearances, and outpatient consultation opinions that are necessitated based on the answers to the screening will be obtained prior to moving forward with the study, as an already established practice within the clinic practice. In addition, any relative contraindications will be further reviewed according to Rossi et al.'s most updated safety guidelines for TMS.

Exclusion Criteria:

* Patients with pre-existing renal disease
* Known allergy to D-serine, or with
* Patients taking medications with known drug-drug interactions
* Children
* Pregnant or breast-feeding women

The investigators will not include children because prior safety and dosing studies excluded children. Although considered safe for TMS, the investigators will not include pregnant or breast-feeding women on the basis of unknown safety profile of exogenous D-serine for these patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire 9 (PHQ-9) | Through TMS treatment course, average of 6-8 weeks; taken at treatment #1, #9, #14, #19, #24, #29, and #34, an average of once per week
  The PHQ-9 is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression. The PHQ-9 test evaluates several factors that revolve around the criteria used to professionally diagnose depression under the current DSM-5. The total score is calculated and can range from zero to 27, with 27 being the highest and indicative of the worst outcome/severity.
  * A score of 20 or higher indicates that severe major depression
  * Scoring between 15 and 19 suggests that there is possibly moderately severe major depression
  * Scoring between 10 and 14 means that you may have a moderate severity depression
  * A score between 5 and 9 reveals that mild symptoms of depression appear to exist

SECONDARY OUTCOMES:
Quick Inventory of Depressive Symptomatology (QIDS SR-16) | Through TMS treatment course, average of 6-8 weeks; taken at treatment #1, #9, #14, #19, #24, #29, and #34, an average of once per week
  This scale is a self-report measure of depression. Questions in the QIDS - SR-116 correlate with the nine DSM-IV symptom criterion domains, including: Sleep disturbance (initial, middle, and late insomnia or hypersomnia) (Q 1 - 4), Sad mood (Q 5), Decrease/increase in appetite/weight (Q 6 - 9), Concentration (Q 10), Self-criticism (Q 11), Suicidal ideation (Q 12), Interest (Q 13), Energy/fatigue (Q 14), and Psychomotor agitation/retardation (Q 15 - 16). Severity of depression can be judged based on the total score as seen below of lowest to highest score values and their correlating severity. Higher scores indicating a worse outcome.
  1-5 = No depression 6-10 = Mild depression 11-15 = Moderate depression 16-20 = Severe depression 21-27 = Very severe depression
Generalized Anxiety Disorder-7 (GAD-7) | Through TMS treatment course, average of 6-8 weeks; taken at treatment #1, #9, #14, #19, #24, #29, and #34, an average of once per week
  The Generalized Anxiety Disorder - 7 Item Scale (GAD-7) is a self-administered questionnaire designed for screening and measuring the severity of generalized anxiety disorder (GAD). The GAD-7 consists of seven items that respondents rate based on their experiences over the past two weeks, with each item scored from 0 (not at all) to 3 (nearly every day). The cumulative score, ranging from 0 to 21, indicates the severity of GAD symptoms, with higher scores corresponding to greater anxiety levels. This simplicity in administration and interpretation makes the GAD-7 a practical tool for healthcare providers to quickly assess anxiety levels and monitor changes over time.

CONTACTS AND LOCATIONS:
Overall Officials: Kerry Ressler, MD, PhD, Study Director — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
The investigators will not share Individual Participant Data.

REFERENCES:
- [Background] Kantrowitz JT, Malhotra AK, Cornblatt B, Silipo G, Balla A, Suckow RF, D'Souza C, Saksa J, Woods SW, Javitt DC. High dose D-serine in the treatment of schizophrenia. Schizophr Res. 2010 Aug;121(1-3):125-30. doi: 10.1016/j.schres.2010.05.012. Epub 2010 Jun 11. PMID 20541910
- [Background] Sehatpour P, Kreither J, Lopez-Calderon J, Shastry AM, De Baun HM, Martinez A, Javitt DC. Network-level mechanisms underlying effects of transcranial direct current stimulation (tDCS) on visuomotor learning in schizophrenia. Transl Psychiatry. 2023 Nov 23;13(1):360. doi: 10.1038/s41398-023-02656-3. PMID 37993420
- [Background] Rossi S, Antal A, Bestmann S, Bikson M, Brewer C, Brockmoller J, Carpenter LL, Cincotta M, Chen R, Daskalakis JD, Di Lazzaro V, Fox MD, George MS, Gilbert D, Kimiskidis VK, Koch G, Ilmoniemi RJ, Lefaucheur JP, Leocani L, Lisanby SH, Miniussi C, Padberg F, Pascual-Leone A, Paulus W, Peterchev AV, Quartarone A, Rotenberg A, Rothwell J, Rossini PM, Santarnecchi E, Shafi MM, Siebner HR, Ugawa Y, Wassermann EM, Zangen A, Ziemann U, Hallett M; basis of this article began with a Consensus Statement from the IFCN Workshop on "Present, Future of TMS: Safety, Ethical Guidelines", Siena, October 17-20, 2018, updating through April 2020. Safety and recommendations for TMS use in healthy subjects and patient populations, with updates on training, ethical and regulatory issues: Expert Guidelines. Clin Neurophysiol. 2021 Jan;132(1):269-306. doi: 10.1016/j.clinph.2020.10.003. Epub 2020 Oct 24. PMID 33243615